CLINICAL TRIAL: NCT00002340
Title: A Randomized, Open-Label Trial of High Dose Atovaquone Versus Low Dose Atovaquone Versus Aerosolized Pentamidine for Prophylaxis of Pneumocystis Carinii Pneumonia in Patients With HIV Infection Who Are Intolerant of TMP/SMX
Brief Title: A Comparison of Atovaquone and Pentamidine in the Prevention of Pneumocystis Carinii Pneumonia in HIV-Infected Patients Who Cannot Take TMP/SMX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 227B; 230
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-08

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Pneumonia, Pneumocystis carinii; Pentamidine; Antifungal Agents; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; atovaquone
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Atovaquone; Pentamidine

INTERVENTIONS:
Drug: Atovaquone
Drug: Pentamidine isethionate

SUMMARY:
To assess whether high dose or low dose atovaquone suspension is more effective than aerosolized pentamidine as prophylaxis against Pneumocystis carinii pneumonia (PCP) in high-risk HIV-infected patients. To compare the safety of chronic administration of the three regimens in patients with advanced HIV disease. To determine the relationship between steady state atovaquone plasma concentrations and prophylactic efficacy against PCP.

DETAILED DESCRIPTION:
Patients are randomized to receive oral atovaquone at 1 of 2 doses once daily or aerosolized pentamidine once every 4 weeks. Treatment continues until 18 months after the last patient is enrolled. Patients are stratified into primary or secondary prophylaxis strata based on prior occurrence of a PCP episode.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antimicrobial agents not specifically prohibited.

Concurrent Treatment:

Allowed:

* Transfusion.

Patients must have:

* HIV positivity.
* Prior PCP (histologically confirmed) OR documented CD4 count < 200 cells/mm3 OR constitutional symptoms such as thrush or unexplained fever (> 100 F) for 2 or more weeks.
* No current or suspected active PCP, and no signs of active PCP on chest x-ray.
* Prior intolerance to TMP/SMX or other trimethoprim or sulfa-containing regimens.
* Life-expectancy of at least 6 months.

NOTE:

* Pregnant women are eligible at the discretion of the investigator.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Significant psychosis or emotional disorder that would preclude study compliance.
* Severe chronic diarrhea (e.g., > five stools/day) that may negatively affect absorption of oral medication.
* Unable to take oral medication or unable or unwilling to take medication with food.

Concurrent Medication:

Excluded:

* Rifampin.
* Other investigational agents except for drugs available through Treatment INDs or expanded access programs.
* Medications likely to have anti-pneumocystis effect (e.g., dapsone, trimethoprim, pyrimethamine, trimetrexate, other DHFR inhibitors, sulfadiazine, sulfamethoxazole, other sulfonamides, primaquine, clindamycin, and sulfonylureas.
* Corticosteroids in greater than physiologic replacement doses for more than 21 consecutive days.
* Systemic therapy for CNS toxoplasmosis, Kaposi's sarcoma, lymphoma, other active malignancies, or other disease that may decrease life expectancy or confound assessment.

Patients with the following prior conditions are excluded:

* History of severe or intractable intolerance to atovaquone or aerosolized pentamidine.
* Prior hypoglycemia, pancreatitis, arrhythmias, or severe hypotension associated with any form of pentamidine.
* Prior enrollment in this protocol. Active substance abuse that would preclude study compliance.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 615

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Goodgame Med Group, Maitland, Florida
  - Bay Area AIDS Consortium, Tampa, Florida
  - Saint Vincent's Hosp and Med Ctr, New York, New York
  - Holmes Hosp, Cincinnati, Ohio
  - Hampton Roads Med Specialists, Hampton, Virginia

REFERENCES:
- [Background] Chan C, Montaner J, Lefebvre EA, Morey G, Dohn M, McIvor RA, Scott J, Marina R, Caldwell P. Atovaquone suspension compared with aerosolized pentamidine for prevention of Pneumocystis carinii pneumonia in human immunodeficiency virus-infected subjects intolerant of trimethoprim or sulfonamides. J Infect Dis. 1999 Aug;180(2):369-76. doi: 10.1086/314893. PMID 10395851